CLINICAL TRIAL: NCT03012633
Title: Rapid Diagnostic of Hyperfibrinolysis in Liver Transplantation
Acronym: FILYTHO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Alexandre OUATTARA, Head of department of Cardiovascular Anesthesia and Critical care, University Hospital, Bordeaux
Other Study IDs: DC 2016/142
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2016-11

CONDITIONS: Liver Transplantation
Keywords: hyperfibrinolysis, Lysis Timer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Lysis timer — Lysis Timer compared with standard laboratory test to diagnose hyperfibrinolysis during liver transplantation.
  Other Names: Global Fibrinolytic Capacity; GFC test

SUMMARY:
During liver transplantation (LT), hyperfibrinolysis is one of the most important modification of haemostasis. It is associated with t-PA and protein C increased activity. Hyperfibrinolysis is frequent, hardly predictable and associated with major bleeding. The diagnostic of hyperfibrinolysis with standard laboratory tests (euglobulin lysis test, t-PA, PAI-1 and D-dimers dosages) does not provide an answer in a delay compatible with the clinical practice in the operating room.

The "Lysis Timer" is a device developed by Hyphen-Sysmex in collaboration with SD Innovation and Charleroi University Hospital (Belgium). It allows the implementation of the "Global Fibrinolytic Capacity", or GFC test, in a complete system associating i) the reagents for in vitro triggering of the clot and its lysis (contact system activators, t-PA, thrombin and calcium), ii) the signal acquisition by the Lysis Timer (able to convert the analogic signal of the absorbance modifications related to clot formation into a numeric signal) and iii) a dedicated software treating the numeric signal to define clot lysis time.

The GFC test, using t-PA to shorten signal acquisition times, is particularly adapted to the diagnosis of hyperfibrinolysis with PAI-1 collapse, of which LT is an example.

DETAILED DESCRIPTION:
The primary aim of this prospective, monocentric, observational study is to evaluate the Lysis Timer as a rapid diagnostic device for hyperfibrinolysis during liver transplantation. Lysis times provided by this device will be compared to the euglobulin lysis times and to the others parameters of fibrinolysis at the different stages of liver transplantation and more specifically at the anhepatic stage and after graft revascularization.

The secondary aims are to compare the results of the Lysis Timer, the thromboelastogram, the thrombin generation test and the standard laboratory tests in the context of hyperfibrinolysis during liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients benefiting from liver transplantation

Exclusion Criteria:

* age under eighteen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients benefiting from liver transplantation
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
clot lysis time | during the liver transplantation surgery
  clot lysis time obtained quickly with "Lysis Timer "is compared with standard laboratory tests to diagnose hyperfibrinolysis during liver transplantation surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre OUATTARA, MD, PhD, Principal Investigator — head of anesthesia department II
Locations (1):
- BORDEAUX UNIVERSITY HOSPITAL Haut Lévêque, Pessac, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roullet S, Labrouche S, Mouton C, Quinart A, Nouette-Gaulain K, Laurent C, Freyburger G. Lysis Timer: a new sensitive tool to diagnose hyperfibrinolysis in liver transplantation. J Clin Pathol. 2019 Jan;72(1):58-65. doi: 10.1136/jclinpath-2018-205280. Epub 2018 Oct 3. PMID 30282673